CLINICAL TRIAL: NCT00365703
Title: Nasogastric Tube vs. Orogastric Feeding Tube in Preterm Infants: Which is Best?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Hillel Yaffe Medical Center, Hillel Yaffe Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 17/2006-1-HY-CTIL
Record Dates: First submitted 2006-08-15; First posted 2006-08-17 (Estimated); Last update posted 2007-12-19 (Estimated); Status verified 2007-12

CONDITIONS: Infant, Premature
Keywords: Infant, Premature; Tube feeding
MeSH Terms: conditions — Premature Birth | interventions — Intubation, Gastrointestinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Orogastric feeding tube.
  Interventions: Procedure: Feeding tube insertion
- 2 (Experimental): Nasogastric feeding tube.
  Interventions: Procedure: Feeding tube insertion

INTERVENTIONS:
Procedure: Feeding tube insertion — 1. Orogastric feeding tube
  2. Nasogastric feeding tube

SUMMARY:
The purpose of this study is to find out which method (nasogastric vs. orogastric) of feeding tube for premature infants results in earlier only oral feeding.

DETAILED DESCRIPTION:
Preterm infants, even as young as 23 weeks gestational age, can be fed enterally at the first week of life. Coordination of sucking and swallowing, and coordination of both and breathing is necessary for efficient and safe oral feeding, and is not well established before the 35th week gestational age. That is why tube feeding is essential for preterm infants younger than that age.

There is no consensus regarding the best way for the feeding tube, i.e. oral vs. nasal, and whether placing the tube should be continuous or intermittently. Nasogastric tube has been associated with vagal responses. Both tubes may cause gastric perforation.

Development and function of oral feeding has been described. It is known that non-nutritive sucking and early introduction of oral feeding accelerate the transition from tube feeding to oral feeding. It is suggested that the preterm infant may experience a maturational lag in vagal function related to ingestive needs, which may contribute to continued feeding difficulties and may be a measurable marker of subtle neurodevelopmental problems. Both oral and nasal feeding tube may interfere with establishment of efficient oral feeding. The purpose of this study is to see whether there is a difference between oral and nasal tube feeding, regarding the institution of oral feeding.

ELIGIBILITY:
Inclusion Criteria:

* All preterm infants, born during one year, who required tube feeding, and later discharged from neonatal intensive care unit.

Exclusion Criteria:

* Infants who died during hospitalization
* Infants with severe neurologic deficit (e.g. after Sarnat II-III asphyxia, or as a part of a syndrome
* Infants with gastrostomy
* Infants who were transferred to another hospital for any reason (e.g. heart surgery)

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2006-09; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The mean post conceptual age at which the infant is fed orally only. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Erez Nadir, MD, Principal Investigator — Hillel Yaffe medical cenetr, Hadera, Israel
Locations (1):
- Neonatal intensive care unit, Hille Yaffe medical center, Hadera, Hadera, Israel

REFERENCES:
- [Background] Lau C, Smith EO, Schanler RJ. Coordination of suck-swallow and swallow respiration in preterm infants. Acta Paediatr. 2003 Jun;92(6):721-7. PMID 12856985
- [Background] Mizuno K, Ueda A. The maturation and coordination of sucking, swallowing, and respiration in preterm infants. J Pediatr. 2003 Jan;142(1):36-40. doi: 10.1067/mpd.2003.mpd0312. PMID 12520252
- [Background] Shiao SY, Youngblut JM, Anderson GC, DiFiore JM, Martin RJ. Nasogastric tube placement: effects on breathing and sucking in very-low-birth-weight infants. Nurs Res. 1995 Mar-Apr;44(2):82-8. PMID 7892144
- [Background] Haxhija EQ, Rosegger H, Prechtl HF. Vagal response to feeding tube insertion in preterm infants: has the key been found? Early Hum Dev. 1995 Mar 17;41(1):15-25. doi: 10.1016/0378-3782(94)01605-o. PMID 7781566
- [Background] Grunebaum M, Horodniceanu C, Wilunsky E, Reisner S. Iatrogenic transmural perforation of the oesophagus in the preterm infant. Clin Radiol. 1980 May;31(3):257-61. doi: 10.1016/s0009-9260(80)80211-x. PMID 7428263
- [Background] Arvedson JC, Lefton-Greif MA. Anatomy, physiology, and development of feeding. Semin Speech Lang. 1996 Nov;17(4):261-8. doi: 10.1055/s-2008-1064103. PMID 8979310
- [Background] Lau C, Schanler RJ. Oral motor function in the neonate. Clin Perinatol. 1996 Jun;23(2):161-78. PMID 8780899
- [Background] Stevenson RD, Allaire JH. The development of normal feeding and swallowing. Pediatr Clin North Am. 1991 Dec;38(6):1439-53. doi: 10.1016/s0031-3955(16)38229-3. PMID 1945550
- [Background] Pinelli J, Symington A. Non-nutritive sucking for promoting physiologic stability and nutrition in preterm infants. Cochrane Database Syst Rev. 2001;(3):CD001071. doi: 10.1002/14651858.CD001071. PMID 11686975
- [Background] Simpson C, Schanler RJ, Lau C. Early introduction of oral feeding in preterm infants. Pediatrics. 2002 Sep;110(3):517-22. doi: 10.1542/peds.110.3.517. PMID 12205253
- [Background] Fucile S, Gisel E, Lau C. Oral stimulation accelerates the transition from tube to oral feeding in preterm infants. J Pediatr. 2002 Aug;141(2):230-6. doi: 10.1067/mpd.2002.125731. PMID 12183719
- [Background] Suess PE, Alpan G, Dulkerian SJ, Doussard-Roosevelt J, Porges SW, Gewolb IH. Respiratory sinus arrhythmia during feeding: a measure of vagal regulation of metabolism, ingestion, and digestion in preterm infants. Dev Med Child Neurol. 2000 Mar;42(3):169-73. doi: 10.1017/s001216220000030x. PMID 10755456